CLINICAL TRIAL: NCT06544824
Title: Accuracy of Markerless Motion Analysis in Comparison with Optoelectronic Motion Capture System
Brief Title: Accuracy Comparison: Optoelectronic Motion Capture and Markerless System
Acronym: OPR
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: GIP1121
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Children, Adult; Motor Disorders
Keywords: Kinematic; Markerless; OpenPose
MeSH Terms: conditions — Motor Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Healthy subjects: This group includes healthy subjects over 4 years of age; with the ability to walk independently without walking aids and/or orthoses.
  Interventions: Other: Measure gait spatiotemporal parameters and kinematics from optoelectronic system; Other: Measure gait spatiotemporal parameters and kinematics from markerless system
- Subjects with a diagnosis of cerebral palsy and right hemiplegia: This group includes subjects with a diagnosis of cerebral palsy and right hemiplegia over 4 years of age; with the ability to walk independently without walking aids and/or orthoses.
  Interventions: Other: Measure gait spatiotemporal parameters and kinematics from optoelectronic system; Other: Measure gait spatiotemporal parameters and kinematics from markerless system
- Subjects with a diagnosis of cerebral palsy and left hemiplegia: This group includes subjects with a diagnosis of cerebral palsy and left hemiplegia over 4 years of age; with the ability to walk independently without walking aids and/or orthoses.
  Interventions: Other: Measure gait spatiotemporal parameters and kinematics from optoelectronic system; Other: Measure gait spatiotemporal parameters and kinematics from markerless system
- Subjects with a diagnosis of spastic paraparesis: TThis group includes subjects with a diagnosis of spastic paraparesis over 4 years of age; with the ability to walk independently without walking aids and/or orthoses.
  Interventions: Other: Measure gait spatiotemporal parameters and kinematics from optoelectronic system; Other: Measure gait spatiotemporal parameters and kinematics from markerless system

INTERVENTIONS:
Other: Measure gait spatiotemporal parameters and kinematics from optoelectronic system — The raw data acquired from motion capture system were processed with Smart Analyzer software (BTS Bioengineering, Milano, Italy). First, the 3D data were filtered and interpolated in case of missing data for short time. Then spatial-temporal parameters (cycle duration, cadence, gait speed, stance phase, swing phase, double-support phase, stride length and step width) and conventional kinematic parameters of traditional Davis marker-set protocols were computed.
Other: Measure gait spatiotemporal parameters and kinematics from markerless system — The two videos were elaborated using OpenPose that returns a set of 25 2D keypoints coordinates for body pose estimation for each video. Key-points were located in relevant body landmarks and it were used to determine the 2D Cartesian coordinates on the sagittal plane and on the frontal plane. The data calculated with routines were filtered and interpolated in case of missing data. With respect to kinematic parameters, the segment and joint angles were measured from the estimated feature points of each joint. Spatiotemporal gait parameters were calculated using successive heel strike and toe-off events.

SUMMARY:
The purpose of this study was to assess the Openpose reliability to measure kinematics and spatiotemporal gait parameters and to evaluate the minimum technical requirements. This analysis used video and optoelectronic motion capture simultaneously recorded. We assessed more of 20 subject with different motor gait impairments

DETAILED DESCRIPTION:
Marker-based Optical motion tracking is the gold standard in gait analysis, but today, markerless solutions are growing rapidly. Treatment of physical impairments could improve if supported with reliable motion capture. Moreover, the use of markerless technology offers numerous advantages for working with pediatric populations under various conditions. In this paper, we assess the Openpose reliability to measure kinematics and spatiotemporal gait parameters and to evaluate the minimum technical requirements., in a population of children with and without gait impairments. Validating markerless methods can open the way for new motion capture techniques and enhance the accessibility of kinematic measurements and improve the treatment of physical impairments.

ELIGIBILITY:
Inclusion Criteria:

* Age over 4 years;
* Ability to walk independently without walking aids and/or orthoses.

Exclusion Criteria:

* Inability to walk independently and safely for short distances without walking aids and/or orthoses.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study includes subjects who previously underwent a functional motor assessment using the SMART DX 100 system at the IRCCS Eugenio Medea Institute. The sample comprises both healthy individuals and those with walking difficulties, all aged over 4 years.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Absolute Error | Through study completion, an average of 1 year
  Absolute errors were calculated for the kinematics parameters and for each spatiotemporal variable by taking the absolute value after subtracting the values obtained using pose estimation methods from the value measured using markerbased motion capture
intraclass correlation coefficients | Through study completion, an average of 1 year
  To confirm whether the data obtained by OpenPose agreed with the data from the optoelectronic system, investigators calculated the ICCs (two-way mixed effects model, absolute agreement, average measurements) between the spatiotemporal and kinematic data from both systems. The ICC values were interpreted as follows: poor agreement for ICC < 0.5, moderate agreement for values between 0.5 and 0.75, good agreement for values between 0.75 and 0.9, and excellent agreement for values greater than 0.90.
cross-correlation coefficients | Through study completion, an average of 1 year
  The cross-correlation coefficients (CCC) between both systems were used to evaluate the similarity of angles during the gait cycle. The CCC values were interpreted as follows: weak or no coupling for values between -0.3 and 0.3, moderate coupling for values between 0.3 and 0.7 or -0.7 and -0.3, and strong coupling for values greater than 0.7 or less than -0.7.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Andreoni, Principal Investigator — IRCCS E.Medea
Locations (1):
- IRCCS E. Medea, Bosisio Parini, Italy, Italy

IPD SHARING:
Plan to Share IPD: No